CLINICAL TRIAL: NCT05628896
Title: Efficacy of a Preoperative Anaemia Clinic in Patients Undergoing Elective Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Eske Kvanner Aasvang, Clinical Professor, Rigshospitalet, Denmark
Other Study IDs: RH-2043-KB1
Record Dates: First submitted 2022-10-25; First posted 2022-11-29 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2023-03

CONDITIONS: Anemia, Iron-Deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Efficacy of a preoperative anaemia clinic in patients undergoing elective abdominal surgery diagnosed with iron deficieny anaemia

DETAILED DESCRIPTION:
Objective: this study aims to investigate how preoperative intravenous iron treatment affects hemoglobin elevations in patients undergoing elective abdominal surgery diagnosed with iron deficiency anaemia and when treatment should be administrated for optimal effect.

Methods: the study is a prospective, descriptive cohort study, where patients are included from a quality improvement project at The Departments of Abdominal Surgery and the Department of Anesthesia, Centre for Cancer and Organ Disease at Rigshospitalet in Denmark. Patients undergoing elective abdominal surgery will be screened for iron deficiency anaemia 1-4 weeks prior to surgery and patients diagnosed with iron deficiency anaemia will be included. Intravenous iron infusion will be administrated preoperatively and Hb will be measured 1-2 days prior to surgery or on day of surgery. The preparation used is ferric derisomaltose (MonoFer, Pharmacosmos A/S, Holbæk, Denmark) with a max single iron dose of 20 mg/kg. The dose administrated is calculated using patient bodyweight and Hb value and administered ≥30 minutes followed by 30 minutes observation including monitoring with 3-lead ECG and pulsoximitri.

Study results will be sought to be published in an international peer-reviewed journal.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with preoperative iron deficiency anaemia
* All patients receiving preoperative or postoperative intravenous iron infusion
* Patients undergoing elective abdominal surgery

Exclusion Criteria:

* Patients missing Hb values after intravenous iron infusion prior to surgery
* Patients undergoing acute abdominal surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients scheduled for elective abdominal surgery diagnosed with iron deficiency anaemia who received a pre- or postoperative intravenous iron infusion. Patients receiving postoperative intravenous iron infusion will be excluded from the analysis.
Sampling Method: Non-Probability Sample
Enrollment: 764 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Assess the possible change in hemoglobin (Hb) concentration in patients with iron deficiency anaemia undergoing intravenous iron infusion of MonoFer prior to abdominal surgery. | Hb values [mM] from blood samples taken before the preliminary examination and 1-2 days prior to surgery in patients receiving intravenous iron infusion
  Preoperative anaemia is defined as:
  * Hb <8,1 mM for men
  * Hb <7,5 mM for women
  Iron deficiency was defined as TSAT <20%. Iron deficiency anaemia was defined as TSAT <20% with concurrent anaemia.
  Paired Student's t-test will be performed to analyze whether intravenous iron infusion prior to surgery results in a significant increased Hb level at the day of surgery in patients with preoperative iron deficiency anaemia. In case data is not normally distributed, data will be analyzed using Wilcoxon signed rank test.

SECONDARY OUTCOMES:
Assess the ideal time point for administration of preoperative intravenous iron infusion of MonoFer and the effect on Hb concentration | Hb values [mM] from blood samples taken before the preliminary examination and 1-2 days prior to surgery in patients receiving intravenous iron infusion. Number of days between infusion of intravenous MonoFer and day of surgery (up to 3 months)).
  To assess if there is a significant difference in patients receiving iron infusion >2 weeks and <2 weeks preoperatively an Unpaired Students T-test will be performed. A comparison of delta Hb values (±SD) will furthermore be investigated.
  To evaluate whether there is an ideal day of preoperative administration, linear regression and correlation analysis will analyze the correlation between delta Hb values and days between administrated treatment and day of surgery.
  Lastly a multiple linear regression will be performed to analyze potential interaction between delta Hb and:
  1. Age
  2. Severity of anaemia
  3. Preoperative chemotherapy

OTHER OUTCOMES:
Investigate the effect of screening elective patients undergoing abdominal surgery preoperatively to prevent preoperative iron deficiency anaemia. | Number of patients undergoing elective abdominal surgery from June 2020 - August 2022 with iron deficiency anaemia who had not been screened and administrated preoperative intravenous iron infusion.
  Number of patients with iron deficiency anaemia on day of surgery who had been screened and administrated intravenous iron infusion and who had not will be calculated and compared (number and percentages).

CONTACTS AND LOCATIONS:
Overall Officials: Eske Kvanner Aasvang, DMSci, Study Chair — Rigshospitalet, Denmark
Locations (1):
- The Departments of Abdominal Surgery and the Department of Anesthesia, Centre for Cancer and Organ Disease at Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided